CLINICAL TRIAL: NCT04909944
Title: Clinical Performance of the I-gel and the Laryngeal Tube Suction Disposable Supraglottic Airway Devices by Novice Intubators During Manual In-line Neck Stabilization: A Randomized Controlled Trial
Brief Title: Performance of the I-gel and the Laryngeal Tube Suction Disposable by Novice Intubators"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS GAITINI MD, Associate Clinical Professor of Anesthesiology, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0069-21-BNZ
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Anesthesia
Keywords: Supraglottic devices; Airway; Insertion success

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-gel supraglottic device insertion for oxygenation (Experimental): i-gel supraglottic device insertion for oxygenation and ventilation
  Interventions: Device: i-gel Supraglottic insertion
- laryngeal tube suction disposable supraglottic insertion for oxygenation (Experimental): laryngeal tube suction disposable insertion for oxygenation and ventilation
  Interventions: Device: Laryngeal Tube Suction Disposable Supraglottic insertion

INTERVENTIONS:
Device: i-gel Supraglottic insertion — i-gel Supraglottic insertion for oxygenation
  Arms: i-gel supraglottic device insertion for oxygenation
Device: Laryngeal Tube Suction Disposable Supraglottic insertion — Laryngeal Tube Suction Disposable Supraglottic insertion for oxygenation
  Arms: laryngeal tube suction disposable supraglottic insertion for oxygenation

SUMMARY:
Establishing a definitive airway is defined as a tube placed in the trachea with cuff inflated below the vocal cords is the first priority in the airway management of the pre-hospital trauma Studies revealed that the success rate of tracheal intubation in the prehospital setting is suboptimal.

The Advance Trauma Life Support suggested the use of the Supraglottic Airway Devices in managing patients who require an advanced airway adjunct, but in whom intubation has failed.

The Laryngeal Tube Suction Disposable (LTS-D), was introduced as an alternative for managing the difficult airway, initially intended for routine clinical use.

Within recent years, laryngeal tubes have also been reported to be successfully used in emergency airway management.

The i-gel disposable airway is proposed as a new supraglottic airway device (SAD) made of a medical grade thermoplastic elastomer. Its unique design does not need an inflatable cuff.

A randomized controlled trail will be conducted. Participants will insert the both supraglottic airway devices to compare performance of ventilation and oxygenation of the patients.

The insertion will be performed on aged 18-75 year patients, scheduled for elective surgery with general anesthesia. The SAD use in the study will be a single use i-gel size 4, an size 5 and the LTS-D size 4 and the size 5.

For induction of anesthesia, all patients will receive premedication with oral diazepam (10 mg). After 3 min of preoxygenation with an inspired oxygen fraction of 100%, anesthesia will be induced with up to 3mcg/kg fentanyl and 2-3 mg/kg propofol and will be maintained with 70% nitrous oxide/30% oxygen and sevoflurane. Neuromuscular blockade will be obtained with rocuronium. After complete neuromuscular blockade, the study procedure will be initiated. The participant will perform one insertion of i-gel or the LTS-D on the patient while manual in-line stabilization of the neck.

Primary outcome measure - insertion success rate. The primary outcome measure will be success rate of effective insertion of the Supraglottic Airway Devices in the patients with registration of the CO2 (carbon di oxide) curve.

Secondary outcome measure - duration in seconds of the insertion. The duration of the Supraglottic Airway Devices insertion will be defined as the duration time, in seconds, from insertion of the Supraglottic Airway Devices in the lips of the patient until will be correctly positioned in the trachea by the participant.

DETAILED DESCRIPTION:
In the combat setting, airway compromise is the second leading cause of preventable death after hemorrhage. Establishing a definitive airway defined as a tube placed in the trachea with cuff inflated below the vocal cords is the first priority in the airway management of the pre-hospital trauma patient, according to the last edition of the Advanced Trauma Life Support (ATLS) textbook, of the American College of Surgeons. However, studies revealed that the success rate of tracheal intubation in the prehospital setting using direct laryngoscopy, the standard intubation technique) is suboptimal. Possible reasons for the failure in achieving definitive airway in trauma patients are the requirement for in-line stabilization of the neck, and the inexperience of the care providers. The Tactical Combat Casualty Care Guidelines recommend using a supra glottic airway device as an option to assist in securing the airway in tactical evacuation phase of care. The utility of a supraglottic airway device is also recommended by the American College of Surgeons. In a randomized controlled trail in patient, the success of blind intubation did not support the use of tracheal intubation via intubating Laryngeal Tube Suction-Disposable (iLTS-D) by novice intubators. However, this study revealed a high success rate (84.6%) of intubating Laryngeal Tube Suction-Disposable placement in the oropharynx, associated with effective ventilation as confirmed by capnography.

The time to obtain successful iLTS-D placement in the oropharynx was 42 sec, which is 2.5 times shorter than the time to achieve tracheal intubation with Direct Laryngoscopy.

These findings suggest that novice intubators can use a second generation Supraglottic Airway Device as the first airway intervention in trauma patients who require immediate airway management.

The ATLS suggested the use of the Supraglottic Airway Devices (SGAD) in managing patients who require an advanced airway adjunct, but in whom intubation has failed or is unlikely to succeed.

The American Association of Anesthesiology include the use of Supraglottic Airway Device in the control of the airway in cases of difficult intubation Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults included the use of SGAD in the Guidelines of difficult intubation.

The 4th National Audit Project of The Royal College of Anaesthetists and The Difficult Airway Society recommends that all hospitals have second generation Supraglottic Airway Devices available for both routine use and rescue airway management.

These devices play a key role as primary and rescue devices in predicted and unanticipated difficult airway management, by providing both a patent airway for oxygenation and ventilation and a conduit for Tracheal Intubation thereby avoiding the disastrous outcomes of 'cannot intubate, cannot oxygenate' situations.

Recently study reported the effectiveness of initial Laryngeal Tube (LT) insertion vs initial Endotracheal Intubation (ETI) in adults out of Hospital cardiac arrest (OHCA). This study concludes that a strategy of initial LT insertion was associated with significantly greater 72-hour survival compare with a strategy of initial Endotracheal Intubation (ETI).

These findings suggest that LT insertion may be considered as an initial airway management strategy in patients with OHCA.

The laryngeal tube and its derivatives, the laryngeal tube suction, were introduced as an alternative for managing the difficult airway, initially intended for routine clinical use.

Within recent years, laryngeal tubes have also been reported to be successfully used for out-of-hospital and emergency airway management.

Recently study reported the effectiveness of initial Laryngeal Tube (LT) insertion vs initial Endotracheal Intubation (ETI) in adults out of Hospital cardiac arrest (OHCA).This study concludes that a strategy of initial LT insertion was associated with significantly greater 72-hour survival compare with the strategy of initial ETI.

These findings suggest that LT insertion may be considered as an initial airway management strategy in patients with OHCA.

The i-gel disposable airway (Intersurgical Ltd, Workingham, UK) is proposed as a new supraglottic airway device made of a medical grade thermoplastic elastomer. Its unique design does not need an inflatable cuff because the thermoplastic elastomer provides the seal Initial studies have demonstrated that the i-gel can be placed more quickly than conventional laryngeal mask airways, which might play a role in prehospital settings other advantages in ease of training, size and weight, cost, safety, and simplicity of use.

The Tactical Combat Casualty Care ( TCCC) suggested the use of extraglottic airways (EGAs) as an option for airway management in Tactical Field Care.

The TCCC recommends the second-generation supraglottic airway device i-gel as the preferred EGA because its gel-filled cuff makes it simpler to use and avoids the need for cuff inflation and monitoring. If an EGA with an air-filled cuff is used, the cuff pressure must be monitored to avoid over pressurization, especially during Tactical Evacuation Care (TACEVAC) on an aircraft with the accompanying pressure changes.

EGA s play a key role as primary and rescue devices in predicted and unanticipated difficult airway management, by providing both a patent airway for oxygenation and ventilation and a conduit for TI , thereby avoiding the disastrous outcomes of 'cannot intubate, cannot oxygenate' situations.

Study design A randomized controlled trial will be conducted. Participants will perform tracheal intubation using The Laryngeal Tube Suction Disposable and their performance will be compared with the use of i-gel to ventilated and oxygenate the patients.

The study will be conducted at the operating room of a Bnai Zion Medical Center, Haifa, Israel. The study will be approved by the Institutional of Human Ethics Committee , and a written consent will be obtained from all patients.

The study will be registered in the Clinical Trial.gov

Study participants Study participants will be medical interns who will be assigned to the Department of Anesthesiology as part of their one-year internship. Medical interns in Israel receive non-formal training in cardiac life support and trauma life support as part of the medical school curriculum. None of the study participants will have a prior clinical experience with the EGAs. Only subjects who accomplished a Cardiac Advanced Life Support course in their 6th year of medical school and had some experience with intubation will requited.

Study patients The intubations will be performed on aged 18-75 year patients, scheduled for elective surgery with general anesthesia, who will have an American Society of Anesthesiologists physical status of I or II, and will agree to undergo the procedure by a novice intubator, supervised by a senior anesthesiologist. To identify the presence of difficult airway preoperatively, a combination of predictors will be used.

Study instruments The EGA use in the study will be a single use i-gel size 4 for medium adult weight 50-90 Kg. and size 5 for large adult more than 90 Kg. and the Laryngeal Tube Suction Disposable size 4 for patients weight 50-90 Kg and size 5 for patients more than 90 Kg.

Study procedure Patients For induction of anesthesia, all patients will receive premedication with oral diazepam (10 or 20 mg). After 3 min of preoxygenation with an inspired oxygen fraction of 100%, anesthesia will be induced with up to 3mcg/kg fentanyl and 2-3 mg/kg propofol and be maintained with 70% nitrous oxide/30% oxygen and sevoflurane. Neuromuscular blockade will be obtained with rocuronium bromide 0.6 mg/kg.

After confirmation of complete neuromuscular blockade, the study procedure will initiate.

After the surgery, the patients will be transferred to the Post Anesthesia Care Unit.

Participants Participants will be randomly assigned to one of the two groups of the study . When patient will be ready to be anesthetized, the participant will enter the operating room.

The participant will then be asked by the study investigator to independently perform one insertion attempt using the EGA i-gel or the LTS-D on the patient while manual in-line stabilization of the neck will be performed by the study investigator. The study investigators will not intervene with the procedure or provide any consultation or recommendation, and participants will not be allowed to watch others performing the procedure. If a failed insertion of the EGA , the study investigator will perform the intubation using direct laryngoscopy.

Primary outcome measure -insertion EGA success rate The primary outcome measure will be success rate verified by inflating the patient's lungs through the EGA using the anesthetic circuit and by the CO2 capnography monitor tracing curve.

Secondary outcome measure - duration in second of the EGA insertion. The time to achieve successful ventilation via bag-mask ventilation will be defined as the duration of time duration from insertion of the laryngoscope or the EGA between the lips of the patient until identification of capnography curve.

Success of correct placement of i-gel or LTS-D within the oropharynx was verified by the insufflation of the patient lungs and the appearance of the CO2 capnography curve.

ELIGIBILITY:
Inclusion Criteria:

* Patient ASA (American Society Anesthesiologists) guidelines I-II
* non pregnancy

Exclusion Criteria:

* Difficult airway
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Insertion success ratio between supraglottic devices the laryngeal tube suction disposable and the i-gel | 30 seconds
  Comparison of the insertion success in the oropharynx of laryngeal tube suction disposable and the i-gel supraglottic devices, insertion success detected by capnography trace